CLINICAL TRIAL: NCT01039389
Title: Promotion of Coronary Collateral Function by Ivabradine-Induced Bradycardia in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Christian Seiler, MD, Professor and Co-Chairman of Cardiology, Department of Cardiology, University Hospital, CH-3010 Bern, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 237/2008
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stable; Coronary Collaterals; Therapeutic Collateral Promotion; Arteriogenesis; Bradycardia
MeSH Terms: conditions — Coronary Artery Disease; Bradycardia | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collateral promotion; PCI after 6 months (Experimental)
  Interventions: Drug: Ivabradine; Drug: Placebo
- Collateral promotion; PCI at baseline (Experimental)
  Interventions: Drug: Ivabradine; Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — bid administration of 5mg ivabradine (max 7.5mg) aiming to reduce resting heart rate to 60/min
  Other Names: Procoralan, I(f)-inhibitor
Drug: Placebo — bid placebo
  Other Names: Placebo control

SUMMARY:
The purpose of this study in patients with chronic stable coronary artery disease treatable by percutaneous coronary intervention (PCI) is to evaluate the long-term efficacy and safety of the orally taken selective I(f)-inhibitor Ivabradine (Procoralan®, Servier Switzerland) with regard to the promotion of collateral growth.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in industrialized countries. Current therapies for restoration of coronary flow are percutaneous coronary intervention (PCI) or surgical revascularization. However, inherent to them are procedure-related risks and the fact that CAD progression is not prevented. Additionally, up to one fourth of all CAD patients are not amenable to standard revascularization therapies. Thus, there is a need for alternative therapies. Coronary collaterals as natural bypasses are anastomoses without an intervening capillary bed between portions of the same coronary artery or between different coronary arteries. The coronary collateral circulation is prevalent in humans and in CAD the amount of collateral flow is directly related to infarct size, all-cause- and cardiac mortality. Thus, the goal is to promote collateral function in the sense of prophylactic myocardial salvage.

Coronary (collateral) blood flow occurs almost entirely during diastole. Fluid shear stress (FSS) is the driving force in the formation, promotion and maintenance of collaterals (i.e. arteriogenesis). It is the product of blood viscosity and shear rate, the latter being the fluid velocity change between different fluid layers which is related to the fluid velocity at the endothelium. Prolongation of diastole via reduction of resting heart rate (RHR) is naturally equal to extension of shear stress at the endothelium. Bradycardia is likely to be the key factor for augmented collateral function: In several animal models, an inverse relation between heart rate and collateral function was found. We have recently confirmed this finding investigating collateral function measurements in normal coronary arteries of our patient population.

The fact that beta blockers depress contractility and unmask beta-adrenergic coronary vasoconstriction has prompted the development of selective I(f)-inhibitors. To date, ivabradine is the only clinically available specific inhibitor of the pacemaker current in the sinuatrial node (called "funny" current, because of permeability for mixed ions and activation by hyperpolarization instead of depolarization, I(f)). It acts as a pure heart rate lowering agent without affecting blood pressure, myocardial contractility, intra-cardiac conduction, or ventricular repolarization. In contrast to beta blockers or calcium channel blockers, it mimics physiological bradycardia and is therefore appropriate for the purpose of this study. By bradycardization in CAD, ischemia is targeted via reduction of myocardial oxygen demand and increase of oxygen supply without negative inotropic, coronary vasoconstrictive, or metabolic effects. In terms of anti-anginal efficacy, ivabradine has been found to be as effective as atenolol or amlodipine.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. 1- to 3-vessel stable coronary artery disease (CAD)
3. At least 1 stenotic lesion suitable for PCI
4. No Q-wave myocardial infarction in the area undergoing CFI measurement
5. Written informed consent to participate in the study

Exclusion Criteria:

1. Acute coronary syndrome
2. CAD treated best by surgical coronary bypass
3. Indications for BB treatment (heart failure, arrhythmias, <3months post-infarct)
4. RHR <60/min without any treatment
5. Sick sinus syndrome, sinuatrial block or >2nd degree atrio-ventricular block
6. Atrial fibrillation
7. Inherited or acquired long-QT syndrome
8. Indwelling pacemaker
9. Severe hepatic or renal failure (creatinine clearance <15ml/min)
10. Hypersensitivity against ivabradine or adjuvants
11. Pre-menopausal women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Collateral flow index (CFI) | 6 months

SECONDARY OUTCOMES:
Myocardial blood flow (MBF) during hyperemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof., Study Chair — Insel Gruppe AG, University Hospital Bern; Michael Stoller, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Tobias Traupe, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Patel SR, Breall JA, Diver DJ, Gersh BJ, Levy AP. Bradycardia is associated with development of coronary collateral vessels in humans. Coron Artery Dis. 2000 Sep;11(6):467-72. doi: 10.1097/00019501-200009000-00004. PMID 10966132
- [Background] DiFrancesco D, Camm JA. Heart rate lowering by specific and selective I(f) current inhibition with ivabradine: a new therapeutic perspective in cardiovascular disease. Drugs. 2004;64(16):1757-65. doi: 10.2165/00003495-200464160-00003. PMID 15301560
- [Background] Meier P, Gloekler S, de Marchi SF, Indermuehle A, Rutz T, Traupe T, Steck H, Vogel R, Seiler C. Myocardial salvage through coronary collateral growth by granulocyte colony-stimulating factor in chronic coronary artery disease: a controlled randomized trial. Circulation. 2009 Oct 6;120(14):1355-63. doi: 10.1161/CIRCULATIONAHA.109.866269. Epub 2009 Sep 21. PMID 19770393
- [Background] Meier P, Gloekler S, Zbinden R, Beckh S, de Marchi SF, Zbinden S, Wustmann K, Billinger M, Vogel R, Cook S, Wenaweser P, Togni M, Windecker S, Meier B, Seiler C. Beneficial effect of recruitable collaterals: a 10-year follow-up study in patients with stable coronary artery disease undergoing quantitative collateral measurements. Circulation. 2007 Aug 28;116(9):975-83. doi: 10.1161/CIRCULATIONAHA.107.703959. Epub 2007 Aug 6. PMID 17679611
- [Derived] Rimoldi SF, Messerli FH, Cerny D, Gloekler S, Traupe T, Laurent S, Seiler C. Selective Heart Rate Reduction With Ivabradine Increases Central Blood Pressure in Stable Coronary Artery Disease. Hypertension. 2016 Jun;67(6):1205-10. doi: 10.1161/HYPERTENSIONAHA.116.07250. Epub 2016 Apr 18. PMID 27091900
- [Derived] Gloekler S, Traupe T, Stoller M, Schild D, Steck H, Khattab A, Vogel R, Seiler C. The effect of heart rate reduction by ivabradine on collateral function in patients with chronic stable coronary artery disease. Heart. 2014 Jan;100(2):160-6. doi: 10.1136/heartjnl-2013-304880. Epub 2013 Nov 1. PMID 24186565